CLINICAL TRIAL: NCT00736242
Title: Treatment of Chronic Hepatitis C in HIV-infected Patients With PegIntron Pen and Rebetol According to German Law (§ 67 Abs 6 AMG)
Brief Title: Post-marketing Surveillance of HIV-infected Patients With Chronic Hepatitis C Treated With PegIntron Pen and Rebetol (Study P04584)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04584
Record Dates: First submitted 2008-07-30; First posted 2008-08-15 (Estimated); Results first posted 2013-04-08 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Chronic Hepatitis C; Hepatitis C; HIV Infections
Keywords: HIV
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; HIV Infections | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PEG-IFN alfa-2b + RBV: Participants received a combination of PEG-IFN alfa-2b plus RBV according to routine clinical practice and locally-approved product recommendations for a minimum of 12 weeks. No investigational medicinal product was provided by the sponsor.
  Interventions: Biological: PEG-IFN alfa-2b; Drug: RBV

INTERVENTIONS:
Biological: PEG-IFN alfa-2b — Peginterferon alfa-2b administered subcutaneously at a dose 1.5 ug/kg/week, according to the European Medicines Agency (EMEA)-approved labeling
  Other Names: SCH 054031; PegIntron
Drug: RBV — Ribavirin administered at a dose of 800-1200 mg/day (on a weight-basis) according to the EMEA-approved labeling
  Other Names: Rebetol; SCH 018908

SUMMARY:
The objective of the study was to assess the safety and efficacy of peginterferon alfa-2b (PEG-IFN alfa-2b) and ribavirin (RBV) administered to participants coinfected with Human Immunodeficiency Virus (HIV) and Hepatitis C Virus (HCV). Participants were treated by general practitioners in clinical practice as part of the post-marketing surveillance study. The study assessed the rates of eradication of the HCV and the rates of serious adverse events reported with PEG-IFN alfa-2b (1.5 ug/kg/week) and RBV (800-1200 mg/day) in common medical practice in Germany.

DETAILED DESCRIPTION:
In this observational, non-interventional study, the time of enrollment and start of treatment was the sole decision of the physician. No investigational medicinal product was provided by the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age eligible for treatment according to the Summary of Product Characteristics (SmPC)
* Presence of chronic Hepatitis C (with elevated liver enzymes and without decompensation)
* Presence of HCV-RNA and known genotype of the infecting hepatitis C virus
* HIV infection confirmed by positive Enzyme Linked Immunosorbent Assay (ELISA) and Western blot and Cluster of differentiation (CD) 4 cell count >200/mL
* Treatment-naïve
* Platelets ≥ 75,000/mm^3
* Neutrophil counts ≥ 1,500/mm^3
* Thyroid Stimulating Hormone (TSH) must be within normal limits
* Hemoglobin ≥ 10 g/dL (females); ≥ 11 g/dL (males)
* Women of childbearing potential must have a routine pregnancy test performed monthly during treatment and for 7 months thereafter. Sexually active female participants of childbearing potential must be practicing adequate contraception (intrauterine device, oral contraceptives, implanted contraceptives, surgical sterilization, barrier method, or monogamous relationship with a male partner who has had a vasectomy or is using a condom (+ spermicide) during the treatment period and for 7 months after stopping treatment.
* Sexually active male participants must be practicing acceptable methods of contraception (vasectomy, use of condom + spermicide, monogamous relationship with a female partner who practices an acceptable method of contraception) during the treatment period and for 7 months after stopping treatment.

Exclusion Criteria:

* Contraindications according to the European approval and to the SmPC
* Pretreatment of chronic hepatitis C
* Liver decompensation
* Hypersensitivity to the active substance or to any interferons or to any of the excipients
* Pregnant woman
* Women who are breast feeding
* Existence of or history of psychiatric condition, particular depression, suicidal ideation or suicide attempt
* A history of severe pre-existing cardiac disease, including unstable or uncontrolled cardiac disease in the previous six months
* Severe debilitating medical conditions, including participants with chronic renal failure or creatinine clearance < 50 ml/min.
* Autoimmune hepatitis or history of autoimmune disease
* Severe hepatic dysfunction or decompensated cirrhosis of the liver
* Pre-existing thyroid disease unless it can be controlled with conventional therapy
* Epilepsy and/or compromised central nervous system function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects coinfected with HIV and HCV seen in common medical practice by general practitioners and clinical doctors at 30 sites all over Germany.
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2005-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 232 participants enrolled, only 229 patients were included in the Safety Analysis Set and had documented baseline data. Three participants were excluded due to violation of inclusion criteria, violation of exclusion criteria and no application of peginterferon alfa-2b (PEG-IFN alfa-2b).
Groups:
- PEG-IFN Alfa-2b + RBV: Participants received a combination of PEG-IFN alfa-2b plus ribavirin (RBV) according to routine clinical practice and locally-approved product recommendations for a minimum of 12 weeks. No investigational medicinal product was provided by the sponsor.
Period: Overall Study
Arm/Group | PEG-IFN Alfa-2b + RBV
Started | 232
Participants in Safety Analysis Set | 229
Completed | 107
Not Completed | 125

BASELINE CHARACTERISTICS:
Arm/Group | PEG-IFN Alfa-2b + RBV
Number analyzed (Participants) | 229
Age, Customized [Number; unit: participants]
  ≤40 years | 108
  ≥40 years | 119
  Missing Data | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 188

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Virologic Response (SVR)
Description: SVR was defined as undetectable serum Hepatitis C Virus ribonucleic acid (HCV-RNA) at End of Treatment (EOT) and at the End of Follow-up (EOF).
Time Frame: From End of Treatment to 24 weeks post-treatment (up to 72 weeks)
Population: Analysis was performed on all participants in the Efficacy Analysis Set (all participants with HCV-RNA detectable for ≥6 months before the first application of PEG-IFN alfa-2b, Human Immunodeficiency Virus [HIV] co-infection, and who had received any amount of PEG-IFN alfa-2b) with documented visits at EOT or at follow-up 24 weeks after EOT.
Measure: Number; unit: participants
Arm/Group | PEG-IFN Alfa-2b + RBV
Number analyzed (Participants) | 181
participants | 73

2. Secondary Outcome: Number of Participants With Rapid Virologic Response (RVR)
Description: RVR was defined as undetectable serum HCV-RNA at week 4.
Time Frame: At Treatment Week 4
Population: Analysis was performed on all participants in the Efficacy Analysis Set (all participants with HCV-RNA detectable for at least 6 months before the first application of PEG-IFN alfa-2b, HIV co-infection, and who had received any amount of PEG-IFN alfa-2b) with a documented visit at Treatment Week 4
Measure: Number; unit: participants
Arm/Group | PEG-IFN Alfa-2b + RBV
Number analyzed (Participants) | 194
participants | 28

3. Secondary Outcome: Number of Participants With Early Virologic Response (EVR)
Description: EVR was defined as undetectable serum HCV-RNA at week 12 and/or a
  ≥2 log decline in HCV-RNA levels at week 12 from baseline.
Time Frame: From Treatment Week 1 to Treatment Week 12
Population: Analysis was performed on all participants in the Efficacy Analysis Set (all participants with HCV-RNA detectable for at least 6 months before the first application of PEG-IFN alfa-2b, HIV co-infection, and who had received any amount of PEG-IFN alfa-2b) with a documented visit at Treatment Week 12.
Measure: Number; unit: participants
Arm/Group | PEG-IFN Alfa-2b + RBV
Number analyzed (Participants) | 180
participants | 101

4. Secondary Outcome: Participant Study Status at End of Follow-up (EOF)
Description: Participant study status was assessed at the End of Follow-up (defined as 24 weeks after the end of treatment) based on serum levels of HCV-RNA.
  SVR was defined as defined as undetectable serum HCV-RNA at EOT and EOF, Relapse was defined as undetectable HCV-RNA at EOT with detectable HCV-RNA at EOF, and Non-response was defined as a detectable serum HCV-RNA at EOT.
Time Frame: From EOT to EOF (up to 72 weeks)
Population: Analysis was performed on all participants in the Efficacy Analysis Set (all participants with HCV-RNA detectable for at least 6 months before the first application of PEG-IFN alfa-2b, with HIV co-infection, and who had received any amount of PEG-IFN alfa-2b) with documented visits at EOT or at follow-up 24 weeks after EOT.
Measure: Number; unit: participants
Arm/Group | PEG-IFN Alfa-2b + RBV
Number analyzed (Participants) | 181
participants
  Not Evaluable/Not Documented | 16
  SVR | 73
  Relapse | 16
  Non-response | 60
  Lost to Follow-up/Premature Discontinuation | 16

5. Secondary Outcome: Number of Participants With Hepatitis C Virus (HCV)-RNA Negativity During PEG-IFN Alfa-2b/RBV Treatment
Description: HCV-RNA negativity/positivity was documented at baseline in the medical history (anamnesis), and assessed within the laboratory (lab) at baseline and during treatment by Polymerase Chain Reaction (PCR).
  HCV-RNA (+) = HCV-RNA positive, HCV-RNA (-) = HCV-RNA negative, HCV-RNA Missing = HCV-RNA data not documented, not applicable, not known, not examined, or missing.
Time Frame: From the Baseline Visit up to EOF (up to 72 weeks)
Population: Efficacy Analysis Set: all participants with HCV-RNA detectable for at least 6 months before the first application of PEG-IFN alfa-2b, HIV co-infection, and who had received any amount of PEG-IFN alfa-2b.
Measure: Number; unit: participants
Arm/Group | PEG-IFN Alfa-2b + RBV
Number analyzed (Participants) | 203
participants
  Baseline (anamnesis) HCV-RNA (+) [n=203] | 193
  Baseline (anamnesis) HCV-RNA (-) [n=203] | 0
  Baseline (anamnesis) HCV-RNA Missing [n=203] | 10
  Baseline (lab) HCV-RNA (+) [n=197] | 187
  Baseline (lab) HCV-RNA (-) [n=197] | 3
  Baseline (lab) HCV-RNA Missing [n=197] | 7
  Week 2 HCV-RNA (+) [n=200] | 27
  Week 2 HCV-RNA (-) [n=200] | 3
  Week 2 HCV-RNA Missing [n=200] | 170
  Week 4 HCV-RNA (+) [n=194] | 104
  Week 4 HCV-RNA (-) [n=194] | 28
  Week 4 HCV-RNA Missing [n=194] | 62
  Week 6 HCV-RNA (+) [n=168] | 14
  Week 6 HCV-RNA (-) [n=168] | 11
  Week 6 HCV-RNA Missing [n=168] | 143
  Week 8 HCV-RNA (+) [n=185] | 37
  Week 8 HCV-RNA (-) [n=185] | 26
  Week 8 HCV-RNA Missing [n=185] | 122
  Week 12 HCV-RNA (+) [n=180] | 50
  Week 12 HCV-RNA (-) [n=180] | 70
  Week 12 HCV-RNA Missing [n=180] | 60
  Week 18 HCV-RNA (+) [n=153] | 22
  Week 18 HCV-RNA (-) [n=153] | 44
  Week 18 HCV-RNA Missing [n=153] | 87
  Week 24 HCV-RNA (+) [n=142] | 14
  Week 24 HCV-RNA (-) [n=142] | 75
  Week 24 HCV-RNA Missing [n=142] | 53
  Week 30 HCV-RNA (+) [n=93] | 8
  Week 30 HCV-RNA- [n=93] | 37
  Week 30 HCV-RNA Missing [n=93] | 48
  Week 36 HCV-RNA (+) [n=85] | 6
  Week 36 HCV-RNA (-) [n=85] | 45
  Week 36 HCV-RNA Missing [n=85] | 34
  Week 42 HCV-RNA (+) [n=78] | 5
  Week 42 HCV-RNA (-) [n=78] | 28
  Week 42 HCV-RNA Missing [n=78] | 45
  Week 48 HCV-RNA (+) [n=73] | 8
  Week 48 HCV-RNA (-) [n=73] | 52
  Week 48 HCV-RNA Missing [n=73] | 13
  EOF HCV-RNA (+) [n=158] | 61
  EOF HCV-RNA (-) [n=158] | 71
  EOF HCV-RNA Missing [n=158] | 26

6. Secondary Outcome: Number of Participants With Human Immunodeficiency Virus (HIV)-RNA Negativity During PEG-IFN Alfa-2b/RBV Treatment
Description: HIV-RNA negativity/positivity was documented at baseline in the medical history (anamnesis), and assessed within the laboratory (lab) at baseline and during treatment.
  HIV-RNA (+) = HIV-RNA positive, HIV-RNA (-) = HIV-RNA negative, HIV-RNA Missing = HIV-RNA data not documented, not applicable, not known, not examined, or missing
Time Frame: From the Baseline Visit up to EOF (up to 72 weeks)
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | PEG-IFN Alfa-2b + RBV
Number analyzed (Participants) | 203
participants
  Baseline (anamnesis) HIV-RNA (+) [n=203] | 106
  Baseline (anamnesis) HIV-RNA (-) [n=203] | 86
  Baseline (anamnesis) HIV-RNA Missing [n=203] | 11
  Baseline (lab) HIV-RNA (+) [n=197] | 97
  Baseline (lab) HIV-RNA (-) [n=197] | 90
  Baseline (lab) HIV-RNA Missing [n=197] | 10
  Week 4 HIV-RNA (+) [n=194] | 16
  Week 4 HIV-RNA (-) [n=194] | 35
  Week 4 HIV-RNA Missing [n=194] | 143
  Week 12 HIV-RNA (+) [n=180] | 27
  Week 12 HIV-RNA (-) [n=180] | 71
  Week 12 HIV-RNA Missing [n=180] | 82
  Week 24 HIV-RNA (+) [n=142] | 25
  Week 24 HIV-RNA (-) [n=142] | 55
  Week 24 HIV-RNA Missing [n=142] | 62
  Week 48 HCV-RNA+ [n=73] | 19
  Week 48 HIV-RNA (-) [n=73] | 38
  Week 48 HIV-RNA Missing [n=73] | 16
  EOF HIV-RNA (+) [n=158] | 58
  EOF HIV-RNA (-) [n=158] | 72
  EOF HIV-RNA Missing [n=158] | 28

7. Secondary Outcome: Median Cluster of Differentiation 4 (CD4) Cell Count During PEG-IFN Alfa-2b/RBV Treatment
Description: The CD4 helper T cell count was used to assess participant HIV status and was determined in the laboratory at baseline and during the study course.
Time Frame: From the Baseline Visit up to EOF (up to 72 weeks)
Population: Analysis was performed on all participants in the Efficacy Analysis Set (all participants with HCV-RNA detectable for at least 6 months before the first application of PEG-IFN alfa-2b, HIV co-infection, and who had received any amount of PEG-IFN alfa-2b) with data available.
Measure: Median (Full Range); unit: cells/μL
Arm/Group | PEG-IFN Alfa-2b + RBV
Number analyzed (Participants) | 193
cells/μL
  Baseline [n=193] | 495.0 [44.0 to 1861.0]
  Week 4 [n=61] | 410.0 [164.0 to 985.0]
  Week 12 [n=94] | 363.0 [110.0 to 1155.0]
  Week 24 [n=86] | 310.0 [93.0 to 838.0]
  Week 48 [n=58] | 330.0 [118.0 to 790.0]
  EOF [n=138] | 484.5 [82.0 to 1303.0]

8. Secondary Outcome: Number of Participants With A Serious Adverse Event (SAE) During PEG-IFN Alfa-2b/RBV Treatment
Description: An SAE was any adverse drug/biologic/device experience occurring at any dose that resulted in death, was life-threatening (i.e. placed the participant, in the view of the initial reporter, at immediate risk of death from the AE as it occurred), was a persistent or significant disability/incapacity, required in-patient hospitalization, or prolonged hospitalization, or led to a
  congenital anomaly or birth defect.
Time Frame: From First Participant Visit (12/30/2005) up to 30 days after Last Participant Visit (12/31/2011).
Population: Safety Analysis Set: All participants who received any amount of PEG-IFN alfa-2b. If the application of any PEG-IFN alfa-2b was not certain, the participant was considered part of this set. Participants who were not treated with PEG-IFN alfa-2b were also included in this set providing they did not violate any inclusion or exclusion criterion.
Measure: Number; unit: participants
Arm/Group | PEG-IFN Alfa-2b + RBV
Number analyzed (Participants) | 229
participants | 16

ADVERSE EVENTS:
Description: Of 232 participants enrolled, only 229 patients were included in the Safety Analysis Set and had documented baseline data. Three participants were excluded due to 1) violation of inclusion criteria, 2) violation of exclusion criteria and 3) no application of PEG-IFN alfa-2b.
Arm/Group | PEG-IFN Alfa-2b + RBV
Serious Adverse Events (participants affected / at risk) | 16/229
Other Adverse Events (participants affected / at risk) | 39/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG-IFN Alfa-2b + RBV (N=229)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 1 (1)
Haemoglobin Decreased (Investigations) | 2 (2)
Weight Decreased (Investigations) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Disturbance in Attention (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Psychotic Disorder (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG-IFN Alfa-2b + RBV (N=229)
Fatigue (General disorders) | 13 (16)
Headache (Nervous system disorders) | 14 (20)
Depression (Psychiatric disorders) | 12 (12)
Sleep Disorder (Psychiatric disorders) | 14 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other